CLINICAL TRIAL: NCT01607736
Title: Pilot Study of Effects of Virtual Gait Training on Walking Stability in Older Adults
Brief Title: Pilot Study of Virtual Gait Training in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: JBMP-VGTinOA-pilot; EK:113/11 (Other Grant/Funding Number: Velux Foundation Grant Project Number 727)
Record Dates: First submitted 2012-05-16; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Frail Elderly
Keywords: falls; walking; healthy older individuals; virtual gait training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inactive Comparator (No Intervention)
- Virtual Gait Training (Experimental)
  Interventions: Behavioral: Virtual Gait Training

INTERVENTIONS:
Behavioral: Virtual Gait Training — The intervention consisted of 12-minute virtual gait training sessions once daily for a total of 14 weekdays within a three-week period. The intervention video showed walking legs of a 30-year-old woman for female and a 46-year-old man for male participants. The video screen was adjusted in height such that it corresponded to the legs of the standing participant, with a mirror placed above it. Participants began the training session with a circa one minute of concentration on the upcoming intervention. Afterwards, the video was started. Participants were instructed to stand (when necessary, to sit) and observe the video and mirror, and to imagine themselves walking. Training sessions were supervised by a physical therapist who gave additional instructions and comments regarding participants' visual/kinesthetic imagination of themselves performing the observed movement. Verbal and physical reactions during training sessions were documented in written form and sometimes videotaped.
  Arms: Virtual Gait Training

SUMMARY:
Older individuals suffer from falls and fear of falling. The purpose of this study was to determine the effectiveness of a novel virtual gait training on walking performance and fear of falling in older adults, and to evaluate the feasibility of the virtual gait training program. The investigators hypothesize that virtual gait training in older adults over a three week period will both improve gait parameters as measured by a GAITRite® electronic walkway system, and reduce their fear of falling as measured by the Falls Efficacy Scale-International version.

DETAILED DESCRIPTION:
The objectives of this study are to determine the effectiveness of virtual gait training on walking performance and fear of falling in older adults and to evaluate the feasibility of the virtual gait training. This prospective interventional study plans to include twelve residents of senior assisted living facilities in Basel, Switzerland, aged 65 years or older with no severe physical or cognitive disabilities, and who had fallen at least once in the preceding 12 months. Each participant will complete 14 12-minute virtual gait training sessions within a three-week period. Gait parameters will be quantified with the GAITRite® electronic walkway system, and fear of falling evaluated with the Falls Efficacy Scale-International version. The investigators hypothesize that 14 virtual gait training sessions in older adults over a three week period will both improve gait parameters as measured by a GAITRite® electronic walkway system, and reduce their fear of falling as measured by the Falls Efficacy Scale-International version.

ELIGIBILITY:
Inclusion Criteria:

* older than 65 years of age
* fall within last 6 months

Exclusion Criteria:

* cognitive deficits
* physical disability

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
gait speed | Change from baseline in gait speed at 3 weeks
  gait speed measure with GAITRite® electronic walkway system

SECONDARY OUTCOMES:
fear of falling | change from baseline at end of week 3
  total score on Falls Efficacy Scale-International version

CONTACTS AND LOCATIONS:
Overall Officials: Reto W Kressig, MD, Principal Investigator — Dept. of Geriatrics, University Hospital Basel, Basel, Switzerland
Locations (1):
- Mobility Center, Basel, Canton of Basel-City, Switzerland